CLINICAL TRIAL: NCT04329884
Title: Use of Cooled Radiofrequency for the Treatment of Hip Pain Associated With OA of the Hip Compared to Intra-articular Steroid Injections
Brief Title: Use of Cooled Radiofrequency for the Treatment of Hip Pain Associated With Hip OA Compared to Intra-articular Steroid Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Antonia Faustina Chen, Associate Professor of Orthopedic Surgery, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Brigham
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intra-articular corticosteroid injections (Active Comparator): The hip and groin areas will be prepped and draped in the usual sterile fashion with ChloraPrep. Preprocedural vital signs will be performed and will be in the nursing chart for review. Radiology guidance will be used to guide needle placement within the affected hip to administer lidocaine and a corticosteroid intra-articularly.
  Interventions: Drug: intra-articular corticosteroid injection
- Cooled radiofrequency ablation (Active Comparator): The hip and groin areas will be prepped and draped in the usual sterile fashion with ChloraPrep. Preprocedural vital signs will be performed and will be in the nursing chart for review. The HALYARD* COOLIEF* SINERGY* Cooled Radiofrequency Probe (sterile, single use) is inserted through a COOLIEF* SINERGY* Introducer used with fluoroscopy guidance in the AP view to visualize the hip joint and sensory nerve areas over the acetabulum (femoral) and ischium (obturator) where the cooled radiofrequency ablation will be applied to create a focal thermal lesion to encompass and denervate the targeted nerves.
  Interventions: Procedure: Cooled RFA treatment with COOLIEF* device

INTERVENTIONS:
Procedure: Cooled RFA treatment with COOLIEF* device — Patients who are randomized to receive CRFA will be given the treatment by a specialist into the affected hip with OA, and the patient will be followed to determine amount of pain relief and improved hip joint function.
  Other Names: cooled radiofrequency ablation (CRFA)
  Arms: Cooled radiofrequency ablation
Drug: intra-articular corticosteroid injection — Patients who are randomized to receive intra-articular corticosteroid injections will be given the treatment by a specialist into the affected hip with OA, and the patient will be followed to determine amount of pain relief and improved hip joint function.
  Other Names: steroid injection
  Arms: Intra-articular corticosteroid injections

SUMMARY:
This will be a multi-center, prospective, single-blinded randomized clinical trial to investigate the effectiveness of using cooled radiofrequency ablation (CRFA) for the treatment of osteoarthritis (OA) hip pain and function in subjects treated with CRFA compared with standard of care intra-articular steroid injections

DETAILED DESCRIPTION:
This prospective, single-blinded randomized clinical trial investigates the effectiveness of using cooled radiofrequency ablation (CRFA) for the treatment of osteoarthritis (OA) hip pain and function compared with standard of care intra-articular steroid injections. This study also aims to determine if CRFA is more effective at decreasing hip pain from OA after treatment and improving hip function in terms of range of motion and walking mobility when compared to corticosteroid hip injections. The primary outcome of interest is a decrease in visual analog scale (VAS) pain as reported following treatment with either a hip injection or following RFA treatment for patients who are not candidates for total hip arthroplasty (THA). Secondary objectives include physical performance at each follow-up time point including range of motion and 50 ft walk test, Hip disability and Osteoarthritis Outcome Score (HOOS) and PROMIS questionnaires at each follow-up time point, patient satisfaction at 24 weeks after treatment, and the number of subjects requesting additional treatment for hip pain during the follow-up period.

The assessments will be conducted by comparing patients with pain from hip OA who get CRFA treatment versus patients who get a hip corticosteroid injection. The research hypothesis is that CRFA will lead to a greater reduction in pain up to 24 weeks +/- 2 weeks following treatment compared to a hip corticosteroid injection. This may result in patients having greater relief of their hip pain which may improve joint function and quality of life with the availability of a new alternative to treat hip OA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects older than 18 years of age presenting with radiographic evidence of hip OA and demonstrating hip pain for at least 30 days (Radiographic evidence of hip OA is defined as Kellegran-Lawrence grade 2-4)
2. Relief of patients' typical hip pain symptoms after a positive diagnostic nerve block test and eligibility for cooled radiofrequency ablation of these same nerves

Exclusion Criteria:

1. Patients who have received any steroid injection in hip within the last 90 days
2. Individuals who cannot consent for themselves such as children and subjects with impaired decision making
3. Local infection at injection site or active systemic infection
4. Anticoagulation status with inability to discontinue medication for appropriate duration for nerve blocks and CRFA given proximity to major artery. (No anticoagulation contraindications for joint injection)
5. Automated implantable cardioverter defibrillator with inability to utilize magnet for CRFA per treating cardiologist
6. Body habitus does not allow for placement of longest needles and electrodes (approximately 15cm) to successfully administer treatment
7. Allergy or severe renal impairment precluding iodinated contrast or magnevist injection despite standard premedication protocol
8. Negative diagnostic nerve block tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in visual analog scale (VAS) pain by 1.5 points | up to 24 weeks +/- 2 weeks after either a hip injection or following CRFA treatment for hip OA pain.
  VAS Pain score is is scored using a ruler where the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post-surgical patients who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
visual analog scale (VAS) pain scores at each follow-up time point | 4 weeks +/- 2 weeks, 8 weeks +/- 2 weeks, 12 weeks +/- 2 weeks, and 24 weeks +/- 2 weeks following treatment, and 6 months and 1 year after the procedure
  VAS Pain score is is scored using a ruler where the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post-surgical patients who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
Physical performance (hip range of motion) | 4 weeks +/- 2 weeks, 8 weeks +/- 2 weeks, 12 weeks +/- 2 weeks, and 24 weeks +/- 2 weeks following treatment
Physical performance (50 ft walk test) | 4 weeks +/- 2 weeks, 8 weeks +/- 2 weeks, 12 weeks +/- 2 weeks, and 24 weeks +/- 2 weeks following treatment
Hip disability and Osteoarthritis Outcome Score (HOOS) | 4 weeks +/- 2 weeks, 8 weeks +/- 2 weeks, 12 weeks +/- 2 weeks, and 24 weeks +/- 2 weeks following treatment, and 6 months and 1 year after the procedure
  This is a patient reported joint-specific score, which may be useful for assessing changes in hip pathology over time, with or without treatment. Scores range from 0 to 100 with a score of 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 4 weeks +/- 2 weeks, 8 weeks +/- 2 weeks, 12 weeks +/- 2 weeks, and 24 weeks +/- 2 weeks following treatment, and 6 months and 1 year after the procedure
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population.
Patient satisfaction with the study treatment via Likert scale questionnaire | 24 weeks +/- 2 weeks after study treatment
  At the final study visit (week 24+/- 2 weeks), subjects will be asked about their satisfaction with the study treatment via a Likert scale questionnaire. Satisfaction will be measured by the following scale: Very dissatisfied (1), Somewhat dissatisfied (2), Neutral satisfaction (3), Somewhat satisfied (4), and Very satisfied (5). The minimum value will be 1 and the maxim value will be 5. Higher scores are a better outcome, while lower scores are a worse outcome.
Number of subjects requesting additional treatment for hip pain during the follow-up period | 12 weeks after study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oladeji LO, Cook JL. Cooled Radio Frequency Ablation for the Treatment of Osteoarthritis-Related Knee Pain: Evidence, Indications, and Outcomes. J Knee Surg. 2019 Jan;32(1):65-71. doi: 10.1055/s-0038-1675418. Epub 2018 Nov 5. PMID 30396206
- [Result] Davis T, Loudermilk E, DePalma M, Hunter C, Lindley D, Patel N, Choi D, Soloman M, Gupta A, Desai M, Buvanendran A, Kapural L. Prospective, Multicenter, Randomized, Crossover Clinical Trial Comparing the Safety and Effectiveness of Cooled Radiofrequency Ablation With Corticosteroid Injection in the Management of Knee Pain From Osteoarthritis. Reg Anesth Pain Med. 2018 Jan;43(1):84-91. doi: 10.1097/AAP.0000000000000690. PMID 29095245
- [Result] Davis T, Loudermilk E, DePalma M, Hunter C, Lindley DA, Patel N, Choi D, Soloman M, Gupta A, Desai M, Cook E, Kapural L. Twelve-month analgesia and rescue, by cooled radiofrequency ablation treatment of osteoarthritic knee pain: results from a prospective, multicenter, randomized, cross-over trial. Reg Anesth Pain Med. 2019 Feb 16:rapm-2018-100051. doi: 10.1136/rapm-2018-100051. Online ahead of print. PMID 30772821
- [Result] Bellini M, Barbieri M. Cooled radiofrequency system relieves chronic knee osteoarthritis pain: the first case-series. Anaesthesiol Intensive Ther. 2015;47(1):30-3. doi: 10.5603/AIT.2015.0003. PMID 25751290
- [Result] Gupta G, Radhakrishna M, Etheridge P, Besemann M, Finlayson RJ. Radiofrequency denervation of the hip joint for pain management: case report and literature review. US Army Med Dep J. 2014 Apr-Jun:41-51. PMID 24706242
- [Result] Rivera F, Mariconda C, Annaratone G. Percutaneous radiofrequency denervation in patients with contraindications for total hip arthroplasty. Orthopedics. 2012 Mar 7;35(3):e302-5. doi: 10.3928/01477447-20120222-19. PMID 22385437
- [Result] Kapural L, Jolly S, Mantoan J, Badhey H, Ptacek T. Cooled Radiofrequency Neurotomy of the Articular Sensory Branches of the Obturator and Femoral Nerves - Combined Approach Using Fluoroscopy and Ultrasound Guidance: Technical Report, and Observational Study on Safety and Efficacy. Pain Physician. 2018 May;21(3):279-284. PMID 29871372